CLINICAL TRIAL: NCT01077947
Title: Comparing the Value of Functional Anesthetic and Provocative Discography in the Surgical Treatment of Discogenic Pain
Brief Title: Value of Functional Anesthetic and Provocative Discography in the Surgical Treatment of Discogenic Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Internal
Sponsor: Northwestern University (Other)
Collaborators: Medtronic Spine LLC (Industry)
Responsible Party: Khalid Malik, M.D., Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: STU00006921
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Discogenic Pain; Low Back Pain
Keywords: low back pain; spinal fusion; Primarily axial low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional anesthetic discography (Active Comparator): The patients disc levels for surgical treatment will be based exclusively on their Functional anesthetic discography results. The discography will be performed at a maximum of two disc levels. Discs showing the following MRI findings will be considered for discography:
  1. Loss of disc signal intensity on T-2 weighted sagittal MR images.
  2. Loss of disc height on sagittal MR images.
  Patients will be followed-up at 3 weeks, 3 months, 6 months and 1 year after the surgery by research personnel. Patients will be asked to complete questionnaires before their discography and at every follow-up visit.
  Interventions: Procedure: Functional anesthetic discography
- Provocative Discography (Active Comparator): The patients disc levels for surgical treatment will be based exclusively on their Provocative Discography results. The discography will be performed at a maximum of two disc levels. Discs showing the following MRI findings will be considered for discography:
  1. Loss of disc signal intensity on T-2 weighted sagittal MR images.
  2. Loss of disc height on sagittal MR images.
  The control disc, in the case provocative discography group must appear normal on the MRI - must have preserved disc height and central disc signal intensity on T-2 weighted images. The provocative discography will be performed using the standard IASP criteria. The patients will be followed-up at 3 weeks, 3 months, 6 months and 1 year after the surgery.
  Interventions: Procedure: Provocative Discography

INTERVENTIONS:
Procedure: Functional anesthetic discography — Functional anesthetic discography will be performed to diagnose discogenic pain and to correctly identify the disc levels for the surgical treatment. Proper identification for disc levels should improve the overall results of surgery for this condition.
  Arms: Functional anesthetic discography
Procedure: Provocative Discography — Provocative Discography will be performed to diagnose discogenic pain and to correctly identify the disc levels for the surgical treatment. Proper identification for disc levels should improve the overall results of surgery for this condition.
  Arms: Provocative Discography

SUMMARY:
Although discography and spinal imaging techniques, either alone or in combination, are commonly used to diagnose discogenic pain, their exact role in predicting surgical results are poorly defined. Our aim in this study is to compare the ability of Functional anesthetic discography (FAD), and Provocative Discography (PD) to diagnose discogenic pain and to correctly identify the disc levels for the surgical treatment. Proper identification for disc levels should improve the overall results of surgery for this condition. Patients with discogenic pain have better outcomes if the disc levels for the fusion surgery are identified by using FAD compared to similar disc level identification by PD.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 to 65 years.
2. Symptoms of at least 6 months duration.
3. Primarily axial low back pain.
4. At least 6 months of conservative treatment, including, physical therapy, injections, chiropractic etc.
5. Patients with overall pain scores of greater than 6/10 (NRS).
6. Recent (within the past 6 months) lumbar spine MRI showing: disc desiccation and loss of disc height of at least one disc level.

Exclusion Criteria:

1. History of previous spine surgery.
2. MRI changes at more than two disc levels on the recent (within the past 6 months) lumbar spine MRI.
3. Clinical or radiological evidence of significant:

   1. Disc herniation
   2. Spinal Stenosis
   3. Spinal Deformity
   4. Spondylolisthesis
   5. Spinal instability or pars-defect
   6. Facet Syndrome
   7. Sacroiliac Joint Dysfunction
   8. Myofascial Pain Syndrome
   9. Fibromyalgia
4. Current issues of:

   1. Litigation
   2. Disability
   3. Drug addiction or substance abuse
   4. Chronic pain medication abuse
5. Current diagnosis of and medication use for unstable anxiety, depression, and/or behavioral disorders.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Pain | One Year
  Numerical Rating Scale (11-point numerical rating, 0-10, scale of pain intensity)
  Standard Morphine Equivalent intake

SECONDARY OUTCOMES:
Physical functioning | One Year
  Oswestry Disability Index
Quality of Life | One Year
  SF-36 health survey
Patient Satisfaction | One Year
  Patient Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Malik, M.D., Principal Investigator — Department of Anesthesiology, Northwestern University, Feinberg School of Medicine